CLINICAL TRIAL: NCT04586153
Title: A Multicenter, Seamless, Randomized, Third-Party-Blind, Clinical Trial to Evaluate the Safety and Efficacy of Meplazumab in Addition to Standard of Care for the Treatment of COVID-19 in Hospitalized Adults
Brief Title: Study to Assess the Effect of Meplazumab on COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Jiangsu Pacific Meinuoke Bio Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MPZ-II-02
Record Dates: First submitted 2020-10-12; First posted 2020-10-14 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — meplazumab; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Meplzaumb (Experimental): This arm is combined with 3 groups, low dose, middle dose, and high dose. Low dose group: First dose: 0.12 mg/kg - Day 1; second dose: control - Day 8 Middle dose group: First dose: 0.2 mg/kg - Day 1; second dose: 0.2 mg/kg - Day 8 High dose group: First dose: 0.3 mg/kg - Day 1; second dose: 0.3 mg/kg - Day 8
  Interventions: Drug: Meplazumab for Injection
- Placebo (Placebo Comparator): First dose: control - Day 1; second dose: control - Day 8
  Interventions: Drug: Sterile normal saline (0.9%)

INTERVENTIONS:
Drug: Meplazumab for Injection — humanized antibody target CD147
  Arms: Meplzaumb
Drug: Sterile normal saline (0.9%) — Sterile normal saline (0.9%)
  Arms: Placebo

SUMMARY:
This phase2/3 study will be conducted to evaluate the safety and efficacy of Meplazumab in addition to Standard of Care for the treatment of Corona Virus Disease(COVID) 19 in hospitalized adults

DETAILED DESCRIPTION:
1. Rationale:

   Meplazumab is a humanized anti-CD147 immunoglobulin 2 (IgG2) monoclonal antibody which is expected to block the binding of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) spike protein to the human host-cell-expressed CD147, thereby blocking entry of SARS-CoV-2 into human tissue. This expectation is based on in vitro functional studies using Vero E6 cells infected with SARS-CoV-2 that demonstrated effective meplazumab mediated virus gene copy number inhibition upwards of 90% as evaluated by quantitative polymerase chain reaction. Meplazumab may also inhibit COVID-19 associated cytokine storm syndrome based on inhibition of the pro inflammatory factor Cyclophilin A host-cell CD147 interaction.
2. Overall Design:

   This is a multicenter, seamless, randomized, third-party-blind, study to evaluate the safety and efficacy of meplazumab for the treatment of COVID 19 in hospitalized adults (≥18 years). Neither the subject nor the investigator shall be aware of the study drug identity, as the study drug is dispensed by a third party (eg, a pharmacist or nurse).

   Enrollment of subjects will be stopped once the total number of planned subjects have completed the Stage 1 Day 29 visit procedures. Once the interim analysis of Stage 1 study data is complete and the Independent Data Monitoring Committee (IDMC) has recommended the meplazumab dose that is safe and effective to carry forward into Stage 2, the study will resume subject enrollment. A summary of the key Stage 1 interim analysis results will be sent to the relevant Health Authorities involved, if requested.
3. Number of Investigators and Study Centers:

   There will be 15 to 20 Investigators, at 12 to 20 study centers globally, participating in this study.
4. Number of Subjects:

   Subjects will be screened 1 day before randomization. Stage 1: Approximately 168 subjects will be randomized and allocated 1:1:1:1 (42:42:42:42) to receive meplazumab low dose, meplazumab medium dose, meplazumab high dose, or control. An interim analysis will be conducted to select the optimal dose of meplazumab compared with the control group based on response rates of clinical improvement at Day 29.

   Stage 2: 276 more subjects will be randomized and allocated 1:1 (138:138) to receive 0.2mg/kg meplazumab or control. At interim analysis, primary endpoint, sample size calculation for Stage 2 will be re evaluated based on the observed outcomes at Stage 1 and will be capped at 300 subjects total.
5. Treatment Groups and Duration:

Study duration for each subject will be 84±7 days from randomization in each stage.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with laboratory-confirmed SARS CoV 2 infection as determined by PCR or other commercial or public health assay, which is FDA cleared or approved for emergency use (test results must be obtained within 72 hours of Day
* A score of Grade 3 (hospitalized, requiring supplemental oxygen) or Grade 4 (hospitalized, on non-invasive ventilation or high flow oxygen devices) on the 6-point ordinal scale.
* Willingness and ability to comply with study-related procedures and assessments.
* Ability to provide informed consent signed by study subject or legally authorized representative.
* Male and/or female

  a)Male subjects:
* A male subject must agree to use contraception as detailed in Appendix 12.3 of this protocol during the treatment period and for at least 6 months, corresponding to time needed to eliminate study treatment for both genotoxic and teratogenic study treatments, after the last dose of study treatment.

  b)Female subjects:
* A female subject is eligible to participate if she is not pregnant (see Appendix 12.3), not planning to get pregnant in the next 6 months, not breastfeeding, and at least 1 of the following conditions applies:

  i) Not a woman of childbearing potential (WOCBP) as defined in Appendix 12.3. OR ii) A WOCBP who agrees to follow the contraceptive guidance in Appendix 12.3 during the treatment period and for at least 130 days, (5 terminal half lives and, for genotoxic products, an additional 30 days, corresponding to time needed to eliminate study treatment plus 30 days for study treatments with genotoxic potential) after the last dose of study treatment.

Exclusion Criteria:

* Any physical examination findings, laboratory abnormality, and/or history of any illness, that in the study Investigator's judgment, could jeopardize the safety of the subject by their participation in the study.
* Subjects with evidence of critical COVID 19 illness, defined by at least 1 of the following: respiratory failure; shock (defined by systolic blood pressure <90 mm Hg, or diastolic blood pressure <60 mm Hg, or requiring vasopressors); or multi-organ dysfunction/failure.
* Subjects requiring extracorporeal membrane oxygenation (ECMO).
* Stage 4 severe chronic kidney disease or requiring dialysis (ie, estimated glomerular filtration rate(eGFR) mL/min/1.73 m2 < 30).
* Pregnant or breast feeding.
* Anticipated transfer to another hospital which is not a study site within 72 hours.
* Allergy to any study medication.
* Use of anticancer, antitransplant rejection, or immunomodulatory biological drug or kinase inhibitor (eg, tocilizumab, sarilumab) or Janus kinase inhibitors (within 30 days of enrollment or 5 times the half-life [whichever is longer]).
* Chronic glucocorticosteroid use equivalent to daily oral prednisone >10 mg per day (10 mg oral prednisone every other day is allowed).
* Live (live-attenuated) vaccines are not permitted within 2 weeks prior to randomization or during the study treatment and safety follow-up periods.
* Subjects participating in another clinical study. There will be a need for washout with 5 half lives depending on the study treatment or 30 days since any previous study, whichever is longer.
* Total bilirubin (TBL) >2 × upper limit of normal (ULN), or alanine aminotransferase (ALT) >5 × ULN, or aspartate aminotransferase (AST) >5 × ULN, or alkaline phosphatase >5 × ULN.
* Platelet <50×109/L, or hemoglobin <60g/L.
* Glomerular filtration rate <30 milliliter(mL)/min/1.73 m2, or serum creatinine increased by 0.5 mg/dL within 7 days, or oliguria (<400 mL/24 hour), or anuria (<100 mL/24 hour).
* Any physical examination findings, laboratory abnormality, and/or history of any illness, that in the study Investigator's judgment, could jeopardize the safety of the subject by their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-18 (Actual)

PRIMARY OUTCOMES:
Mortality (based on the interim analysis of Stage 1 data) | During the evaluation period (Day 1 to Day 29)
  Mortality (based on the interim analysis of Stage 1 data)
Proportion of subjects alive and discharged without supplemental oxygen | During the evaluation period (Day 1 to Day 29)
  To evaluate live discharge

SECONDARY OUTCOMES:
Changes from baseline in cytokine, chemokines and related inflammatory factors. | During the evaluation period (Day 1 to Day 29)
  To evaluate pharmacodynamic (PD) response to administration of meplazumab, including cytokine, chemokines and related inflammatory factors (IL-2、IL-4、IL-6、IL-7、IL-8、IL-10、IL-12p70、IL-15、IL-17A、IL-1RA、IL-2Rα、MCP-1、MIP-1β、IP-10、TNFα、IFN-γ).
Viral load | During the evaluation period (Day 1 to Day 29)
  Changes from baseline in viral load. Viral load will be determined by qPCR for COVID-19 in nasopharyngeal swab.
Viral negative rate of SARS-Cov-2 nucleic acid | During the evaluation period (Day 1 to Day 29)
  Viral negative rate of SARS-Cov-2 nucleic acid.

CONTACTS AND LOCATIONS:
Locations (1):
- Pesquisare Saúde, Santo André, São Paulo, Brazil

REFERENCES:
- [Derived] Bian H, Chen L, Zheng ZH, Sun XX, Geng JJ, Chen R, Wang K, Yang X, Chen SR, Chen SY, Xie RH, Zhang K, Miao JL, Jia JF, Tang H, Liu SS, Shi HW, Yang Y, Chen XC, Malhotra V, Nasir N, Khanum I, Mahmood F, Hamid S, Stadnik CMB, Itinose K, de Oliveira CCC, Dusilek C, Rivabem L, Cavalcante AJW, Lopes SS, Saporito WF, Fucci FJC, Simon-Campos JA, Wang L, Liu LN, Wang QY, Wei D, Zhang Z, Chen ZN, Zhu P. Meplazumab in hospitalized adults with severe COVID-19 (DEFLECT): a multicenter, seamless phase 2/3, randomized, third-party double-blind clinical trial. Signal Transduct Target Ther. 2023 Jan 30;8(1):46. doi: 10.1038/s41392-023-01323-9. PMID 36717539
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343